CLINICAL TRIAL: NCT03740087
Title: Search for the Transfer of Bovine miRNA to Humans by Comparing the Omnivore Group With a Vegan Group After a Dietary Intervention
Brief Title: Search for Bovine miRNA Transference to Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, Cristina Rodriguez-Padilla, Principal Investigator, Universidad Autonoma de Nuevo Leon
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Bovine miRNA assay FCB
Record Dates: First submitted 2018-11-06; First posted 2018-11-14 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Vegan Diet
Keywords: miRNA; Xenomirs; Diet; Vegan
MeSH Terms: interventions — Diet, Vegan

STUDY DESIGN:
Intervention Model Description: Baseline blood samples were obtained after 12 hours overnight fast; the postprandial miRNA state was measured after intake of a meal with beef (test meal) that consisted of 200 g roast beef with salad (lettuce, tomato, lentils) and a cup of rice. The control diet consisted of the same intervention, without the roast beef. Each intervention day the meals were prepared with fresh food. Participants ate meals under control of the study staff. Postprandial samples were collected at 2, 4 and 6 hours after the diet intervention. The subjects did not eat or drink again until the end of sample collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omnivorous diet (Experimental): This group was assigned a meal containing beef (test meal) that consisted of 200 g roast beef with salad (lettuce, tomato, lentils) and a cup of rice.
  Interventions: Other: Omnivorous diet
- Vegan diet (Active Comparator): This group was assigned a control meal consisted of salad (lettuce, tomato, lentils) and a cup of rice.
  Interventions: Other: Vegan diet

INTERVENTIONS:
Other: Omnivorous diet — Determine if the transfer of bovine miRNAs is carried out after a meal containing beef.
  Arms: Omnivorous diet
Other: Vegan diet — Used as a baseline for miRNA levels in blood
  Arms: Vegan diet

SUMMARY:
Background: Foods derived from plants and animals contain miRNAs, and, some reports have detected diet-derived miRNAs circulating in mammalian serum. It is still unclear if the miRNAs present in food can be absorbed by the gastrointestinal tract and brought to the tissues to perform regulatory functions. The transfer of functional exogenous miRNA has been demonstrated in bacterial and viral infections but it is less well characterized in mammals. Edible bovine tissues contain unique profiles of human-homologous miRNAs that withstand cooking. If miRNAs from other species can cross the gastrointestinal barrier, it could have implications in gene regulation and health.

Objective: Determine whether miRNAs from beef cross the gastrointestinal barrier and are transferred to human plasma.

Methods: The investigators obtained fasting plasma from 29 healthy subjects divided in two groups: the omnivore group (6 men, 8 women) and the vegan group (8 men, 7 women; control group). Each participant was given a standard meal with or without beef depending on their group, then the plasma was collected at 2, 4 and 6 hours after the meal. The changes in the levels of of miR-1, miR-10b, miR-22, miR-92 and miR-192 were analysed by quantitative Polymerase Chain Reaction (qPCR).

DETAILED DESCRIPTION:
Diet plays an important role in both health and disease processes; the study of the influence of diet on the expression and regulation of genes will allow a greater understanding of the relationship between diet and health. One of the most studied gene regulation mechanisms at present is that of microRNAs (miRNAs). miRNAs are small noncoding RNA (approximately ~22 nucleotides) that regulate gene expression at the post-transcriptional level and influence processes such as development, homeostasis, immune response, metabolism and epigenetic processes. miRNAs bind to specific sequences in target mRNA transcripts to repress translation or induce mRNA degradation. miRNAs are stably present in different biofluids and some can be directly taken up by recipient cells for control of gene expression and cellular functions.

The transfer of functional exogenous RNA has been demonstrated in bacterial and viral infections but it is less well characterized in mammals. Foods derived from plants and animals contain miRNAs, and, some reports have detected diet-derived miRNAs circulating in mammalian serum. These findings support cross-kingdom transfer of specific miRNAs to mammalian tissue after food consumption. However, it's still unclear if miRNAs present in food derived from plants and animals can be absorbed by the gastrointestinal tract and brought to the tissues to perform regulatory functions for the cross regulation of gene expression between species. Delivering functional miRNAs from diet-derived sources across the gastrointestinal barrier could be relevant for nutrition, agriculture, human health and could have many potential applications in therapeutic targeting. In light of the controversial findings on diet-derived miRNAs, the question must be examined to determine the transfer of functional exogenous miRNA in mammals. The investigators studied the possible transfer of diet-derived miRNAs from animal tissue to human plasma because beef is an important diet component in Northeastern Mexico, and its consumption has been associated as a potential risk factor for different pathologies, including colorectal cancer.

Methods Study participants: The protocol was approved by an ethical committee. Thirty volunteers, fifteen omnivorous and fifteen vegans (control group), were enrolled in the study. One omnivore subject did not complete the trial. Written informed consent was obtained from all participants prior to enrollment in the study. To verify the health status of the participants, anthropometric measures, hematic biometry and serum chemistry were performed.

Inclusion and exclusion criteria: Healthy volunteers ages 18 to 30 years, able to provide informed consent, with similar anthropometric characteristics were recruited. The participants were divided in two groups: omnivorous and vegan (control). Inclusion criteria for omnivorous subjects was that they should consume beef at least three times per week. The inclusion criteria for vegan subjects was that they should have followed a strict vegan diet for at least one year. Exclusion criteria for all subjects included pregnancy, menstruation during study sample collection, use of medicine or food supplements, intestinal malabsorption and intolerance to ingredients included in the diet intervention.

Study procedure: Baseline blood samples were obtained after 12 hours overnight fast; the postprandial miRNA state was measured after intake of a meal with beef (test meal) that consisted of 200 g roast beef with salad (lettuce, tomato, lentils) and a cup of rice. The control diet consisted of the same intervention, without the roast beef. Each intervention day the meals were prepared with fresh food. Participants ate meals under control of the study staff. Postprandial samples were collected at 2, 4 and 6 hours after the diet intervention. The subjects did not eat or drink again until the end of sample collection.

Human plasma blood samples were collected into vacuum tubes containing EDTA; approximately 5 mL of blood was collected according to standard procedures at each time point (0, 2, 4 and 6 hours). Plasma was separated by centrifugation for 15 minutes at 2,000 × g at room temperature followed by freezing at -80 °C until analyses were performed.

RNAs isolation: Plasma RNA extraction: thawed plasma samples were centrifuged and plasma supernatant (200 µL) was used for purifying total RNA including small RNAs; RNA extraction was carried out using the miRNeasy Serum/Plasma Kit (Qiagen) according to the manufacturer's instructions.

Beef RNA extraction: Total RNA including small RNAs was extracted from raw and cooked beef using miRNeasy Mini Kit (Qiagen) following the manufacturer's instructions. Samples of 50 mg flash-frozen raw or cooked beef were placed into 700µL lysis reagent for disruption and homogenization immediately using the PRO200 homogenizer (PRO Scientific). The RNA was eluted in 30 µl RNase-free water. Quantity and purity were determined using a Nanodrop ND-1000.

qRT-PCR assay: The quantification of the miRNAs 1, 10b, 22, 92a and 192 was performed as shown: 4 µL of total RNA were used as a template for miRNA reverse transcription. Reverse transcription was performed using the Universal cDNA synthesis kit, (Exiqon): 0.5 µL of synthetic miRNA SPIKE (UniSp6) was added to each sample for normalization of miRNA plasma levels. Real-time qPCR was performed by using the ExiLENT SYBR® Green PCR Master Mix and primers miRCURY LNA Universal RT microRNA PCR, (Exiqon) for hsa-miR-1-3p, hsa-miR-10b-5p, hsa-miR-22-3p, hsa-miR-192-5p and hsa-miR-92a-3p. The PCR program and the dissociation curve analysis were carried out in a LightCycler Nano thermal cycler (Roche) under the conditions described by the manufacturer.

The relative quantification method was validated and the miRNA quantification in the omnivore group was carried out using the method 2-ΔΔCt, the normalizer used was the Spike in UniSp6 and the calibrator was the average value ΔCt of the control group at each time point (0, 2, 4 and 6 hours). Spike in UniSp6 was used as normalizer because of the lack of endogenous controls established for normalization in serum and plasma samples. Each sample was analyzed in triplicate including the Spike in UniSp6 and the negative controls. Data was obtained data for the quantitative miRNA detection in plasma after a meal with beef compared with the control group (vegan meal).

Data analysis: The miRNAs normal distribution was determined by the Kolmogorov-Smirnov test. Descriptive statistics were performed with the 2-ΔΔCt values of both study groups at each collection times (0, 2, 4 and 6 h). miRNAs differential detection between the omnivore and the control group was evaluated by t-student test at different postprandial time points was compared to fasting detection using the ANOVA test. Pearson correlations were performed to associate the miRNAs levels with a control or omnivorous diet. The analysis was done with the use of IBM SPSS Statistics 20 and differences were considered significant if p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* For omnivorous subjects was that they should consume beef at least three times per week.
* For vegan subjects was that they should have followed a strict vegan diet for at least one year

Exclusion Criteria:

* For all subjects included pregnancy, menstruation during study sample collection, use of medicine or food supplements, intestinal malabsorption and intolerance to ingredients included in the diet intervention.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2015-04-13 (Actual); Primary Completion 2015-11-16 (Actual); Study Completion 2016-05-22 (Actual)

PRIMARY OUTCOMES:
Relative amount of miR-1, miR-10b, miR-22, miR-92 and miR-192 in plasma | Change from Baseline microRNA levels at 2, 4 and 6 hours after intervention
  Quantification of miR-1, miR-10b, miR-22, miR-92 and miR-192 in plasma after meal time

CONTACTS AND LOCATIONS:
Overall Officials: Fermín Mar-Aguilar, Dr., Principal Investigator — Universidad Autonoma de Nuevo Leon
Locations (1):
- Cristina Rodriguez-Padilla, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palmer JD, Soule BP, Simone BA, Zaorsky NG, Jin L, Simone NL. MicroRNA expression altered by diet: can food be medicinal? Ageing Res Rev. 2014 Sep;17:16-24. doi: 10.1016/j.arr.2014.04.005. Epub 2014 May 14. PMID 24833329
- [Background] Kim VN. MicroRNA biogenesis: coordinated cropping and dicing. Nat Rev Mol Cell Biol. 2005 May;6(5):376-85. doi: 10.1038/nrm1644. PMID 15852042
- [Background] Kim VN, Han J, Siomi MC. Biogenesis of small RNAs in animals. Nat Rev Mol Cell Biol. 2009 Feb;10(2):126-39. doi: 10.1038/nrm2632. PMID 19165215
- [Background] Krol J, Loedige I, Filipowicz W. The widespread regulation of microRNA biogenesis, function and decay. Nat Rev Genet. 2010 Sep;11(9):597-610. doi: 10.1038/nrg2843. Epub 2010 Jul 27. PMID 20661255
- [Background] Kroh EM, Parkin RK, Mitchell PS, Tewari M. Analysis of circulating microRNA biomarkers in plasma and serum using quantitative reverse transcription-PCR (qRT-PCR). Methods. 2010 Apr;50(4):298-301. doi: 10.1016/j.ymeth.2010.01.032. Epub 2010 Feb 8. PMID 20146939
- [Background] Kosaka N, Izumi H, Sekine K, Ochiya T. microRNA as a new immune-regulatory agent in breast milk. Silence. 2010 Mar 1;1(1):7. doi: 10.1186/1758-907X-1-7. PMID 20226005
- [Background] Kuwabara Y, Ono K, Horie T, Nishi H, Nagao K, Kinoshita M, Watanabe S, Baba O, Kojima Y, Shizuta S, Imai M, Tamura T, Kita T, Kimura T. Increased microRNA-1 and microRNA-133a levels in serum of patients with cardiovascular disease indicate myocardial damage. Circ Cardiovasc Genet. 2011 Aug 1;4(4):446-54. doi: 10.1161/CIRCGENETICS.110.958975. Epub 2011 Jun 2. PMID 21642241
- [Background] Zhang L, Hou D, Chen X, Li D, Zhu L, Zhang Y, Li J, Bian Z, Liang X, Cai X, Yin Y, Wang C, Zhang T, Zhu D, Zhang D, Xu J, Chen Q, Ba Y, Liu J, Wang Q, Chen J, Wang J, Wang M, Zhang Q, Zhang J, Zen K, Zhang CY. Exogenous plant MIR168a specifically targets mammalian LDLRAP1: evidence of cross-kingdom regulation by microRNA. Cell Res. 2012 Jan;22(1):107-26. doi: 10.1038/cr.2011.158. Epub 2011 Sep 20. PMID 21931358
- [Background] Baier SR, Nguyen C, Xie F, Wood JR, Zempleni J. MicroRNAs are absorbed in biologically meaningful amounts from nutritionally relevant doses of cow milk and affect gene expression in peripheral blood mononuclear cells, HEK-293 kidney cell cultures, and mouse livers. J Nutr. 2014 Oct;144(10):1495-500. doi: 10.3945/jn.114.196436. Epub 2014 Aug 13. PMID 25122645
- [Background] Yang J, Farmer LM, Agyekum AA, Elbaz-Younes I, Hirschi KD. Detection of an Abundant Plant-Based Small RNA in Healthy Consumers. PLoS One. 2015 Sep 3;10(9):e0137516. doi: 10.1371/journal.pone.0137516. eCollection 2015. PMID 26335106
- [Background] Dickinson B, Zhang Y, Petrick JS, Heck G, Ivashuta S, Marshall WS. Lack of detectable oral bioavailability of plant microRNAs after feeding in mice. Nat Biotechnol. 2013 Nov;31(11):965-7. doi: 10.1038/nbt.2737. No abstract available. PMID 24213763
- [Background] Snow JW, Hale AE, Isaacs SK, Baggish AL, Chan SY. Ineffective delivery of diet-derived microRNAs to recipient animal organisms. RNA Biol. 2013 Jul;10(7):1107-16. doi: 10.4161/rna.24909. Epub 2013 May 3. PMID 23669076
- [Background] Witwer KW, McAlexander MA, Queen SE, Adams RJ. Real-time quantitative PCR and droplet digital PCR for plant miRNAs in mammalian blood provide little evidence for general uptake of dietary miRNAs: limited evidence for general uptake of dietary plant xenomiRs. RNA Biol. 2013 Jul;10(7):1080-6. doi: 10.4161/rna.25246. Epub 2013 Jun 3. PMID 23770773
- [Background] Chan SY, Snow JW. Formidable challenges to the notion of biologically important roles for dietary small RNAs in ingesting mammals. Genes Nutr. 2017 Jul 7;12:13. doi: 10.1186/s12263-017-0561-7. eCollection 2017. PMID 29308096
- [Background] Humphreys KJ, Conlon MA, Young GP, Topping DL, Hu Y, Winter JM, Bird AR, Cobiac L, Kennedy NA, Michael MZ, Le Leu RK. Dietary manipulation of oncogenic microRNA expression in human rectal mucosa: a randomized trial. Cancer Prev Res (Phila). 2014 Aug;7(8):786-95. doi: 10.1158/1940-6207.CAPR-14-0053. PMID 25092886
- [Background] Papaioannou MD, Koufaris C, Gooderham NJ. The cooked meat-derived mammary carcinogen 2-amino-1-methyl-6-phenylimidazo[4,5-b]pyridine (PhIP) elicits estrogenic-like microRNA responses in breast cancer cells. Toxicol Lett. 2014 Aug 17;229(1):9-16. doi: 10.1016/j.toxlet.2014.05.021. Epub 2014 May 28. PMID 24877718
- [Background] Huggett JF, Foy CA, Benes V, Emslie K, Garson JA, Haynes R, Hellemans J, Kubista M, Mueller RD, Nolan T, Pfaffl MW, Shipley GL, Vandesompele J, Wittwer CT, Bustin SA. The digital MIQE guidelines: Minimum Information for Publication of Quantitative Digital PCR Experiments. Clin Chem. 2013 Jun;59(6):892-902. doi: 10.1373/clinchem.2013.206375. Epub 2013 Apr 9. PMID 23570709
- [Background] Schmittgen TD, Livak KJ. Analyzing real-time PCR data by the comparative C(T) method. Nat Protoc. 2008;3(6):1101-8. doi: 10.1038/nprot.2008.73. PMID 18546601
- See also: Cottrill, KA, Stephen C, Y. Diet-Derived MicroRNAs: Separating the Dream from Reality. microRNA Diagnostics and Therapeutics; 2014. p. 46-57. — https://www.ingentaconnect.com/content/doaj/20846843/2014/00000001/00000001/art00001